CLINICAL TRIAL: NCT03256617
Title: The Development of a Cognitive Reassurance Training Program and Its Impact on Physical Therapist and Patient Outcomes
Brief Title: The Development of a Cognitive Reassurance Training Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting beyond September 10, 2018 would mean that the training occurred more than a year in the past. For this reason, we terminated recruitment.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jake Magel, Research Assistant Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 00100188
Record Dates: First submitted 2017-08-08; First posted 2017-08-22 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Low Back Pain
Keywords: low back pain; cognitive reassurance; physical therapist training
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Pre-post test design for the therapists followed by a prospective cohort of patients.
  We anticipate 50 physical therapy providers and 150 patients for a total of 200 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Provider training (Experimental)
  Interventions: Other: Cognitive reassurance training

INTERVENTIONS:
Other: Cognitive reassurance training — The 2-day training program includes 3 sessions that will consist of interactive didactic lectures, solving case studies and role-playing activities. The first session uses lecture and cases to present models of pain and disability, evidence based predictors of disability and delayed recovery and evidence based interventions for patients with low back pain. The second session uses role playing and case studies help the providers to 1) develop skills in identifying maladaptive beliefs about pain in patients with low back pain and 2) develop the skills to address diagnostic uncertainty and negative pain beliefs and 3) develop skills to educate patients with low back pain. The third session will use role playing and case studies to refine the provider' skills in providing cognitive reassurance to patients with low back pain.

SUMMARY:
The focus of this proposal is to evaluate the feasibility of a cognitive reassurance training program by examining changes in physical therapist low back pain beliefs and skills with training and evaluating the quality with which physical therapists apply cognitive reassurance to patients. The secondary focus is to examine the association between physical therapist application of cognitive reassurance and short-term changes in patients' low back pain beliefs and expectations.

DETAILED DESCRIPTION:
Identifying strategies to favorably alter unhelpful cognitions of patients with recent onset low back pain is a research priority and could help curb the transition from acute to chronic low back pain; lessening the need for prolonged and costly management. Current evidence suggests that psychological factors, including maladaptive pain beliefs and avoidant behaviors and expectations for recovery, are associated with poor outcomes in patients with low back pain. Recently, considerable attention has been given to training non-psychologists to provide psychologically based interventions for patients with low back pian. A recent review of interventions that included psychological approaches noted that all of the trials that failed to show beneﬁt included delivery of the intervention by non-psychologists. Authors suggest that increasing the effort in selecting, training, supervising and assessing the competence of the practitioners delivering the treatment could improve results.

Low back pain comprises approximately 50% of the caseload of outpatient physical therapists physical therapists making physical therapists ideally positioned to manage the unhelpful cognitions of patients with low back pain. However, physical therapists often feel unprepared when managing the cognitive factors associated with low back pain. The purpose of this project is to develop and assess the effectiveness of a training program for physical therapists that focuses on cognitive reassurance; a novel cognitive intervention for patients with low back pain.

Cognitive reassurance is a communication approach in which maladaptive beliefs and expectations are identified. Tailored explanations for the patient's conditions are then provided, possible prognosis and treatment are discussed, and clariﬁcations are offered. With adequate training, physical therapists could utilize cognitive reassurance to promote patients' understanding of his/her condition and modify maladaptive low back pain-related beliefs and expectations.

The proposed pilot study will use a pre-post design to examine the impact of cognitive reassurance training on the low back pain beliefs and skills in physical therapists and physical therapist assistants. Following the training the investigators will recruit patients who have scheduled an evaluation for low back pain with the physical therapists who attended the training. Patient data will be collected at baseline before the evaluation and follow up data at 2, 4 and 8 weeks.

The specific aims are: 1) Evaluate the feasibility of a cognitive reassurance training program for physical therapists that focuses on modifying physical therapists' beliefs and improving physical therapists' skill in the application of cognitive reassurance for patients with acute/subacute low back pain. 2) Evaluate the application of cognitive reassurance by physical therapists to patients with acute/sub-acute low back pain. 3) Examine the association between physical therapist application of cognitive reassurance and short-term changes in the patient's low back pain beliefs and expectations (low back pain beliefs, self-efficacy, pain catastrophizing, fear-avoidance).

ELIGIBILITY:
Therapist inclusion criteria:

* University of Utah Health Care physical therapists and physical therapist assistants
* Employed at least 20 hours a week
* Licensed in the state of Utah

Therapist exclusion criteria:

* None

Patient inclusion criteria

* Primary reason for scheduling an evaluation with a physical therapist is low back pain (defined as symptoms of pain and/or numbness between the 12th rib and buttocks with or without referral in to one or both legs
* Current episode of low back pain ≤ 12 weeks duration
* Age 18-64
* Ability to read and speak English

Patient exclusion criteria

* Report being referred to physical therapy for specific low back pathology (e.g. fracture)
* Any lumbar surgery in the past 6 months
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Change in back beliefs questionnaire for health care providers | Baseline, 5 days
  Measures providers' beliefs about back pain pre and post training
Low back pain vignettes | End of 2nd day of therapist training
  Measures provider decision making related to cognitive reassurance
Skills assessment | End of 2nd day of therapist training
  Assess skills in the provision of cognitive reassurance during role-playing activity

SECONDARY OUTCOMES:
Change in the Pain Catastrophizing Scale | Baseline, 4 weeks and 8 weeks
  Measure of patient's pain catastrophizing
Change in fear the Avoidance Beliefs Questionnaire | Baseline, 4 weeks and 8 weeks
  Measure of patient's fear-avoidance beliefs.
Change in the Pain Self-efficacy Questionnaire | Baseline, 4 weeks and 8 weeks
  Measure of patient's pain self-efficacy
Change in the Back Beliefs Questionnaire | Baseline, 4 weeks and 8 weeks
  Measure of patient's back beliefs
Patient check list | 2 weeks following initial evaluation for low back pain by a physical therapist
  Measure whether key messages of cognitive reassurance were perceived by the patient.
Open-ended question | 2 weeks following the initial evaluation for low back pain by a physical therapist
  Asks the patient to list the most important things they learned learned in physical therapy
Provider check list | 2 weeks status post initial evaluation of patient with low back pain
  Measures whether key cognitive reassurance messages were provided to the patient by the provider

CONTACTS AND LOCATIONS:
Overall Officials: Jake S Magel, PT, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Care Out Patient Physical Therapy Clinics, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No